CLINICAL TRIAL: NCT04435171
Title: Comparison of Postoperative Early Period Quality of Life of Patients With Open and Robot Assisted Kidney Transplantation: a Prospective Observational Study
Brief Title: Comparison of Postoperative Early Period Quality of Life of Patients With Open and Robot Assisted Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Renal Transplantation
Record Dates: First submitted 2020-05-22; First posted 2020-06-17 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Quality of Life
Keywords: End Stage Renal Disease; Renal Transplantation; Quality of Life
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open renal transplantation: Patients who were performed open renal transplantation due to end stage renal disease.
  Interventions: Procedure: Renal transplantation
- robot assisted renal transplantation: Patients who were performed robot assisted renal transplantation due to end stage renal disease
  Interventions: Procedure: Renal transplantation

INTERVENTIONS:
Procedure: Renal transplantation — Open or robot assisted renal transplantation

SUMMARY:
The investigators aimed to investigate the quality of life in patients with end-stage renal disease who underwent open or robot-assisted renal transplantation. Also, the investigators sought to determine the parameters which can affect the quality of life in these patients

DETAILED DESCRIPTION:
Patients who underwent open or robot-assisted renal transplantation at Bakirkoy Sadi Konuk Training and Research Hospital between June 2016 and December 2018 constituted the target population of this study. After application of the inclusion and exclusion criteria, the patient group was divided into two groups as per the surgical technique (i.e., open vs. robot-assisted). Demographic data, preoperative and postoperative data of all patients were collected prospectively. The quality of life of the patients was assessed preoperatively and on the postoperative 30th day

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75
* Who were diagnosed with End Stage Renal Disease (i.e., estimated glomerular filtration rate loer than 20 ml/minute or symptomatic uremia or dialysis requirement)
* Received a kidney from a live donor

Exclusion Criteria:

* Patients with mental retardation, dementia, and psychotic or cognitive disorders, including delirium
* Patients who underwent deceased renal transplantation and who underwent simple bilateral nephrectomy or any other surgical procedure concurrent with Open renal transplantation
* Patients who died or had graft failure during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were performed open or robot assisted renal transplantation due to End Stage Renal Disease
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Percentage of change for Quality of Life (measure : Short Form 36) after open and robot assisted renal transplantation | From just before the treatment and up to 30 days after the surgery was performed
  Percentage of change for quality of life (measure : Short Form 36) for patients who performed open and robot assisted renal transplantation due to end stage renal disease. Scores of the Short Form-36 Health Survey vary between 0 and 100, a score of 0 corresponds to the lowest quality, while 100 indicates the highest quality.

CONTACTS AND LOCATIONS:
Overall Officials: Mithat Ekşi, Principal Investigator — Bakırkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakirkoy Dr Sadi Konuk Training and Research Hospital, Department of Urology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No